CLINICAL TRIAL: NCT02885779
Title: Comparison of 2 Techniques of Invasive Mini Surgery: Coelioscopy Mini-trocar and Monotrocar in the Adnexa no Carcinologic Surgery : Forward-looking Observational Study.
Acronym: ANTATROC
Status: Completed | Type: Observational
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: ANTATROC-IPC 2015-011
Record Dates: First submitted 2016-08-18; First posted 2016-09-01 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Gynecologic Surgical Procedures for Adnexa Surgery in Ovarian Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient having an operating indication of adnexa surgery: Patient having an operating indication of adnexa surgery : unilateral or bilateral adnexectomy

SUMMARY:
The advantages of the celioscopy mini--trocar and monotrocar technical are recognized.

There is however no forward-looking or retrospective study comparing the microcomputed-celioscopy (use of microphone) - trocar of 3mm of diameter in access celioscopic pluri--trocar) in the celioscopy monotrocar ( a single intra-umbilical section) in gynecological surgery.

The objective of this preliminary study is to compare both surgical care in terms of morbidity died operating, in adnexa surgeries.

ELIGIBILITY:
Inclusion Criteria :

* Age > 18 ans
* OMS = 2
* Patient having an operating indication of adnexa surgery : unilateral or bilateral adnexectomy

Exclusion Criteria:

* Contraindication to coelioscopy intervention

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Operating indication of adnexa surgery : unilateral or bilateral adnexectomy
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2015-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Immediate post operative pains | Up to 1 month
  consumption of analgesic for pains in immediate operating comment
Court term post operative pains | Up to 2 month
  consumption of analgesic for pains
Medium term post operative pains | Up to 3 month
  consumption of analgesic for pains

SECONDARY OUTCOMES:
Complications per operating | During surgery
  Blood loss
Complications per operating | During surgery
  Addition of trocar
Complications post operating | Up to 1 month
  Duration of hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Paoli-Calmettes, Marseille, Bouches-du-Rhône, France

IPD SHARING:
Plan to Share IPD: No